CLINICAL TRIAL: NCT02250742
Title: The Effect of Dry Needling on Trunk Muscle Function in Low Back Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Gali Dar, PhD, researcher, University of Haifa
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 045/11
Record Dates: First submitted 2014-07-13; First posted 2014-09-26 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Low Back Pain
Keywords: ultrasound imaging; acupuncture; back muscles; spine; muscle strength
MeSH Terms: conditions — Low Back Pain | interventions — Dry Needling; Acupuncture Therapy

ARMS (2):
- low back pain group (Experimental): Dry needling to the lumbar multifidus muscles using a deep insertion technique with 4 needles (2 on each side of the spine) will be utielized. The needles will be left in situ for 10 minutes.
  Interventions: Other: dry needling
- healthy group (Active Comparator): Dry needling to the lumbar multifidus muscles using a deep insertion technique with 4 needles (2 on each side of the spine) will be utilized. The needles will be left in situ for 10 minutes.
  Interventions: Other: dry needling

INTERVENTIONS:
Other: dry needling — Dry needling uses traditional acupuncture needles without injecting any liquid. Dry needling is based on traditional Western medicine whereby the needle insertion sites are located in known anatomical landmarks such as skeletal muscles, fascia and occasionally joints, tendons and bone/tendon junctions.
  Other Names: acupuncture

SUMMARY:
The study will establish data on the function of trunk muscles in healthy and low back pain patient's pre and post dry needling treatment. This will help in understanding the underlying mechanism of this treatment and reveal the effect of dry needling on muscle performance.

Study hypothesis is that an improvement of back muscle function following dry needling procedure will be found.

DETAILED DESCRIPTION:
Dry needling of muscles is mainly used for the management of pain in musculoskeletal disorders. Yet, the association between dry needling and motor performance of muscles is still unclear.

This study aims to investigate the immediate effect of dry needling on lumbar multifidus muscles' function in healthy and low back pain subjects.

The sample will be divided into: low back pain group and control (healthy) group. Both groups will receive dry needling to the lumbar multifidus muscles using a deep insertion technique with 4 needles (2 on each side of the spine). The needles will be left in situ for 10 minutes. Ultrasound imaging will be used to measure multifidus muscles' thickness, pre and post- procedure during rest in a prone position and during contralateral active straight leg extension.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-60 years.
* Healthy individuals or individuals with main complaint of low back pain (LBP)

Exclusion Criteria:

* Patients with "red flags" for a serious spinal condition, for example: tumor, compression fractures, infection, cancer.
* Signs of nerve root compression (positive straight leg raise <45 degrees, decreased reflexes, decrease sensation or decreased strength in the lower extremities).
* Pregnancy.
* Previous surgery to the lumbar spine
* History of congenital lumbar or pelvic anomalies
* Physical therapy for LBP was provided in the 6 months prior to participation in the study
* Patients who are unable to lie prone for 30 minutes.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in Multifidus muscle thickness | baseline and Immediately after dry needling procedure at the same session
  Multifidus muscle thickness will be measured using diagnostic ultrasound imaging

CONTACTS AND LOCATIONS:
Overall Officials: Gali Dar, PhD, Principal Investigator — University of Haifa, Department of Physical Therapy
Locations (1):
- University of Haifa, Haifa, Israel